CLINICAL TRIAL: NCT03377504
Title: Clinical Evaluation of the Effects of Mirror Therapy in Patients With Complex Regional Pain Syndrome (CRPS) Type 1:Prospective Randomized Single Blind Controlled Study
Brief Title: Clinical Evaluation of the Effects of Mirror Therapy in Patients With Complex Regional Pain Syndrome (CRPS) Type 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Ayşe A Küçükdeveci, MD, Professor of Physical Medicine and Rehabilitation, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03-109-17
Record Dates: First submitted 2017-12-14; First posted 2017-12-19 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Complex Regional Pain Syndrome Type I
Keywords: complex regional pain syndrome; mirror therapy; rehabilitation
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: Prospective randomized single blind controlled study
Who Masked: Outcomes Assessor
Masking Description: single blind (outcomes assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mirror group (Experimental): Routine physical therapy and exercise program will be applied to all patients for a total of 4 weeks, 5 days a week, 1 hour/day. Mirror therapy will be applied to the mirror group for 30 minutes per day in addition to this routine treatment.
  Interventions: Behavioral: mirror therapy
- control group (Active Comparator): Routine physical therapy and exercise program will be applied to all patients for a total of 4 weeks, 5 days a week, 1 hour/day. A total of 20 sessions of treatment will be given to each patient.
  Interventions: Behavioral: Routine physical therapy and exercise program

INTERVENTIONS:
Behavioral: mirror therapy — Mirror therapy will include wrist flexion/extension, ulnar/radial deviation, hand finger flexion/extension and abduction/adduction, thumb abduction/adduction/opposition, and forearm supination/pronation movements as well as various object grasping activities according to the status of the patient's hand functions.
  Arms: mirror group
Behavioral: Routine physical therapy and exercise program — Routine physical therapy and exercise program including contrast baths, hot pack, TENS, desensitization, exercises and occupational therapy will be applied to all patients
  Arms: control group

SUMMARY:
CRPS Type 1 can occur after traumas, surgical applications or central nervous system disorders. The triggering factor in CRPS type 1 is fracture in about half of the cases. Mirror therapy is an innovative treatment approach that is cheap, easy to administer and non-invasive. It is thought that this treatment may be complementary to other rehabilitation methods.Neurophysiologic effects of mirror therapy are noted in the brain, especially in the parietal region, cerebellum, basal ganglia and premotor cortex. Mirror therapy is also effective through the mirror neuron system. Mirror therapy triggers neuroplasticity by increasing the connection between neurons in the brain and thereby enhances communication between the motor and the sensory cortex. Recent studies have shown the positive effects of mirror therapy in patients with CRPS Type 1 disease. There are two randomized controlled trials showing the efficacy of mirror therapy in patients with CRPS Type 1 after stroke. Only one pilot study was performed in patients with CRPS Type 1 who were traumatic origin. There are no randomized controlled trials investigating the efficacy of mirror therapy in CRPS Type 1 patients who developed secondary to trauma in the literature. The purpose of this study is to investigate the clinical effects of mirror therapy applied in addition to routine rehabilitation program in patients with traumatic CRPS Type 1. The investigators hypothesized that adjunctive mirror therapy to classical rehabilitation program would result in better outcomes compared with the classical program only.

DETAILED DESCRIPTION:
This study is planned as a prospective randomized single blind controlled study. It was approved by the Ankara University Faculty of Medicine Ethics Committee and was conducted in accordance with the Declaration of Helsinki. This study will include 36 patients with CRPS type 1 who are referred to the Depart-ment of Physical Medicine and Rehabilitation, Hand Rehabilitation Unit at the Medical Faculty of Ankara University. Patients included in the scope of the study will randomly be divided into 2 groups as mirror group and control group. Random allocation software (RAS) program will be used to assign the patients to the treatment groups with "block randomization" method and to create the randomization scheme. In this single blinded study, all patients will be evaluated by the same physician (Dr. Elif Can Ozdemir). The physician will be blind to patient's assignment. Routine physical therapy and exercise program including contrast baths, hot pack, transcutaneous electrical nerve stimulation (TENS), desensitization, exercises and occupational therapy will be applied to all patients for a total of 4 weeks, 5 days a week, 1 hour/day. Mirror therapy will be applied to the mirror group for 30 minutes per day in addition to this routine treatment. Mirror therapy will include wrist flexion/extension, ulnar/radial deviation, hand finger flexion/extension and ab-duction/adduction, thumb abduction/adduction/opposition, and forearm supina-tion/pronation movements as well as various object grasping activities according to the status of the patient's hand functions. A total of 20 sessions of treatment will be given to each patient. The therapy will be given by the physiotherapists in the Hand Rehabilitation Unit. All individuals participating in the study will be assessed before and immediately after the treatment and also 1 month at follow-up. Each assessment will include pain severity, grip strength, lateral pinch strength, hand circumference measurements, hand dexterity, hand function in daily living activities, and health-related quality of life.As the primary outcome variable, the difference in pain measured by the Numerical Rating Scale between baseline and post-treatment is based. In the mirror group, at least 1 point difference in pain according to the control group is evaluated by Mann Whitney U test and it is necessary to take a total of 36 patients with 81% power and 5% error in each group, assuming 1 as the group standard deviation. Mann Whitney U and Wilcoxon test are planned for paired samples. P value of less than .05 is considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals over 18 years of age
* CRPS type 1 diagnosis according to 2003 Budapest diagnostic criteria
* Patients who developed CRPS Type 1 due to traumatic causes (surgical procedures, fractures, immobilization)
* Patients who agree to participate in the study and sign the informed consent form

Exclusion Criteria:

* Patients with peripheral nerve injuries (those with a diagnosis of CRPS type 2 according to Budapest criteria)
* Patients with CRPS Type 1 after central nervous system injury (stroke)
* Patients in the acute and post-acute rehabilitation who have had primary or secondary tendon repair of the hand
* The presence of comorbid conditions (e.g. decompensated heart failure, chronic renal insufficiency, malignancy) that would impair the functioning of the person and the health-related quality of life
* The presence of comorbid disease affecting hand function (e.g. rheumatoid arthritis, psoriatic arthritis or other inflammatory diseases that cause hand involvement)
* Patients with acute deep venous thrombosis and arterial thrombosis of the upper extremity
* Patients with arterial / venous injury and / or undergoing arterial revascularization
* Patients with excessive alcohol and inappropriate opioid use
* Patients with untreated psychiatric problems (major depression, anxiety, schizophrenia, etc.)
* Patients with recurrent CRPS Type 1

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Pain severity | change from baseline at 4 weeks and 8 weeks
  "0-10 Numeric Rating Scale (NRS)" will be used to assess current pain severity. 0 points minimum 10 points indicates the maximum value. Low scores are associated with better clinical outcomes.

SECONDARY OUTCOMES:
Grip strength | change from baseline at 4 weeks and 8 weeks
  The Jamar dynamometer will be used to measure the grip strength. The best result of the 3 sequential measurements will be taken into account
Lateral pinch strength | change from baseline at 4 weeks and 8 weeks
  A pinchmeter will be used to measure the lateral pinch strength. The best result of the 3 sequential measurements will be taken into account.
Hand circumference measurements | change from baseline at 4 weeks and 8 weeks
  Two measurements will be made: one at the level of ulnar styloid process, second at the level of the third distal metacarpal tip
Hand dexterity | change from baseline at 4 weeks and 8 weeks
  Moberg pick up test will be used.
Hand function in daily living activities | change from baseline at 4 weeks and 8 weeks
  Cochin Hand Function Scale (CHFS) will be used.0 points minimum 90 points shows the maximum value. Low scores are associated with better clinical outcomes.
Health-related quality of life | change from baseline at 4 weeks and 8 weeks
  The Nottingham Health Profile (NHP) will be used

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Adile Küçükdeveci, Principal Investigator — Ankara University
Locations (1):
- Ankara University Faculty of Medicine, İbn-i Sina Research and Application Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwenkreis P, Maier C, Tegenthoff M. Functional imaging of central nervous system involvement in complex regional pain syndrome. AJNR Am J Neuroradiol. 2009 Aug;30(7):1279-84. doi: 10.3174/ajnr.A1630. Epub 2009 Apr 22. PMID 19386737
- [Background] Maihofner C, Seifert F, Markovic K. Complex regional pain syndromes: new pathophysiological concepts and therapies. Eur J Neurol. 2010 May;17(5):649-60. doi: 10.1111/j.1468-1331.2010.02947.x. Epub 2010 Feb 18. PMID 20180838
- [Background] Swart CM, Stins JF, Beek PJ. Cortical changes in complex regional pain syndrome (CRPS). Eur J Pain. 2009 Oct;13(9):902-7. doi: 10.1016/j.ejpain.2008.11.010. Epub 2008 Dec 19. PMID 19101181
- [Background] Ramachandran VS, Rogers-Ramachandran D. Synaesthesia in phantom limbs induced with mirrors. Proc Biol Sci. 1996 Apr 22;263(1369):377-86. doi: 10.1098/rspb.1996.0058. PMID 8637922
- [Background] Sutbeyaz S, Yavuzer G, Sezer N, Koseoglu BF. Mirror therapy enhances lower-extremity motor recovery and motor functioning after stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2007 May;88(5):555-9. doi: 10.1016/j.apmr.2007.02.034. PMID 17466722
- [Background] Stevens JA, Stoykov ME. Using motor imagery in the rehabilitation of hemiparesis. Arch Phys Med Rehabil. 2003 Jul;84(7):1090-2. doi: 10.1016/s0003-9993(03)00042-x. PMID 12881842
- [Background] Samuelkamaleshkumar S, Reethajanetsureka S, Pauljebaraj P, Benshamir B, Padankatti SM, David JA. Mirror therapy enhances motor performance in the paretic upper limb after stroke: a pilot randomized controlled trial. Arch Phys Med Rehabil. 2014 Nov;95(11):2000-5. doi: 10.1016/j.apmr.2014.06.020. Epub 2014 Jul 23. PMID 25064777
- [Background] Dohle C, Pullen J, Nakaten A, Kust J, Rietz C, Karbe H. Mirror therapy promotes recovery from severe hemiparesis: a randomized controlled trial. Neurorehabil Neural Repair. 2009 Mar-Apr;23(3):209-17. doi: 10.1177/1545968308324786. Epub 2008 Dec 12. PMID 19074686
- [Background] Cacchio A, De Blasis E, De Blasis V, Santilli V, Spacca G. Mirror therapy in complex regional pain syndrome type 1 of the upper limb in stroke patients. Neurorehabil Neural Repair. 2009 Oct;23(8):792-9. doi: 10.1177/1545968309335977. Epub 2009 May 22. PMID 19465507
- [Background] Moseley GL. Graded motor imagery for pathologic pain: a randomized controlled trial. Neurology. 2006 Dec 26;67(12):2129-34. doi: 10.1212/01.wnl.0000249112.56935.32. Epub 2006 Nov 2. PMID 17082465
- [Background] Giraux P, Sirigu A. Illusory movements of the paralyzed limb restore motor cortex activity. Neuroimage. 2003 Nov;20 Suppl 1:S107-11. doi: 10.1016/j.neuroimage.2003.09.024. PMID 14597303
- [Background] Moseley LG, Gallace A, Spence C. Is mirror therapy all it is cracked up to be? Current evidence and future directions. Pain. 2008 Aug 15;138(1):7-10. doi: 10.1016/j.pain.2008.06.026. Epub 2008 Jul 14. No abstract available. PMID 18621484
- [Background] Rizzolatti G, Craighero L. The mirror-neuron system. Annu Rev Neurosci. 2004;27:169-92. doi: 10.1146/annurev.neuro.27.070203.144230. PMID 15217330
- [Background] McCabe CS, Haigh RC, Ring EF, Halligan PW, Wall PD, Blake DR. A controlled pilot study of the utility of mirror visual feedback in the treatment of complex regional pain syndrome (type 1). Rheumatology (Oxford). 2003 Jan;42(1):97-101. doi: 10.1093/rheumatology/keg041. PMID 12509620
- [Background] Pervane Vural S, Nakipoglu Yuzer GF, Sezgin Ozcan D, Demir Ozbudak S, Ozgirgin N. Effects of Mirror Therapy in Stroke Patients With Complex Regional Pain Syndrome Type 1: A Randomized Controlled Study. Arch Phys Med Rehabil. 2016 Apr;97(4):575-581. doi: 10.1016/j.apmr.2015.12.008. Epub 2015 Dec 23. PMID 26723854
- [Background] Garry MI, Loftus A, Summers JJ. Mirror, mirror on the wall: viewing a mirror reflection of unilateral hand movements facilitates ipsilateral M1 excitability. Exp Brain Res. 2005 May;163(1):118-22. doi: 10.1007/s00221-005-2226-9. Epub 2005 Mar 8. PMID 15754176
- [Background] Yavuzer G, Selles R, Sezer N, Sutbeyaz S, Bussmann JB, Koseoglu F, Atay MB, Stam HJ. Mirror therapy improves hand function in subacute stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2008 Mar;89(3):393-8. doi: 10.1016/j.apmr.2007.08.162. PMID 18295613
- [Background] Wasner G, Schattschneider J, Binder A, Baron R. Complex regional pain syndrome--diagnostic, mechanisms, CNS involvement and therapy. Spinal Cord. 2003 Feb;41(2):61-75. doi: 10.1038/sj.sc.3101404. PMID 12595868